CLINICAL TRIAL: NCT05783934
Title: Evaluation of the Degree of Demyelination and Remyelination in Multiple Sclerosis (MS) Detected by Brain Positron Emission Tomography With Amyloid Markers (PET-CT 18F-Florbetaben) and Comparison With MRI Findings
Brief Title: Demyelination and Remyelination in Multiple Sclerosis (MS) Detected by Brain Amyloid PET-CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CE 2585
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: MRI; 18F-Florbetaben PET/CT
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-Florbetaben PET/CT scan (Experimental): All the partecipants will undergo PET/CT scan evaluation after 18F-florbetaben administration
  Interventions: Diagnostic Test: 18F-florbetaben PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-florbetaben PET/CT — The PET/CT study will be performed using a dual time acquisition protocol consisting of an early acquisition and a late acquisition.
  Early acquisition Early acquisition starts with the patient already positioned on the PET/CT bed and venous access available.
  A low-dose CT scan is performed for attenuation correction, the PET acquisition is started in list mode and a couple of seconds after the start, 300 MBq of 18F-Florbetaben is administered followed by washing with 10 ml of saline.
  Early acquisition will last 30 minutes. Late acquisition A low-dose CT scan is performed to correct for attenuation and anatomical localisation, followed by a 20-minute list mode PET acquisition so that images are acquired after 90 minutes (tolerance: +10 minutes) of radiopharmaceutical uptake.

SUMMARY:
The goal of this clinical trial study is to evaluate the presence of relationships between PET and MRI images indicative of chronic inflammatory activity (smoldering plaques), apparent absence of inflammatory activity (silent plaques without microglial rim), or indicative of more recent inflammatory activity, in contrast-enhanced areas or in T2/Flair-positive areas of not distant onset in patients diagnosed with progressive (secondary or primary) stage multiple sclerosis and in patients in relapse and remission.

Laboratory analysis of serum markers will be performed: neuronal and glial cytoskeletal proteins (e.g., Nf-L, pN-FH, GFAP), and the levels of neurotrophic factors (e.g., BDNF, GDNF) and cytokines (e.g., TNFα, IL-6, IL-1β, interferon) will be evaluated.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune disease affecting the central nervous system with consequent onset of various sensory, motor, sphincter and sometimes cognitive symptoms. It is characterised by the presence of lympho-monocytic inflammatory infiltrates, demyelination, axonal damage, activation of innate immunity, astrogliosis and remyelination. In the last few years, Magnetic Resonance Imaging (MRI) has made enormous progress in the diagnosis and follow-up of patients, highlighting encephalic and spinal lesions, their number and relative lesion burden, location and cortical involvement as well as the presence of blood-brain barrier alterations in the earliest stages of the disease, associated with the activation of acquired immunity with subsequent inflammatory damage.

The demyelination plaques have on their outer edge a thin wall of iron-containing microglial cells that can be detected by high-resolution magnetic susceptibility MRI sequences and techniques. Such plaques, known by neuropathologists as 'smoldering' plaques, are characterised by a concentrically widening periphery causing myelin and neuronal damage while in the centre of the lesion the process of myelin loss becomes complete. Smoldering plaques, more frequent in progressive forms of the disease, are peculiar of MS compared to other demyelinating diseases and are associated with a negative prognostic significance.

Positron Emission Tomography (PET) is a technique that allows to analyze the in vivo metabolism of certain components of the central nervous system, such as neurons and glia, and, in particular cases, to highlight synaptic function and abnormal protein accumulations. In recent years, PET has been used in MS especially for research purposes: it allows to assess the degree of demyelination and remyelination by using amyloid tracers that bind to the white substance, as well as the degree of microglial activation or synaptic impairment applying particular tracer radio isotopes (TPSO ligands or the glycoprotein 2A of synaptic vesicles). The combination of MRI and PET could provide detailed information not only on the degree and extent of the nervous system impairment, but also on the most affected cell populations, on the metabolic activity of the affected encephalic areas and on the degree of success of the damage repair attempts.

The aim of this research project is to study, applying MRI and PET techniques, a population of progressive MS patients (PMS) with a relatively significant impairment and a population of patients with a relapsing-remitting form of the disease (RRMS) with a less significant neurological impairment. The purpose is to study chronically active or 'smoldering' plaques, with magnetic susceptibility MRI techniques and PET techniques with amyloid tracers, chronically inactive plaques and more recent T2/Flair positive plaques, with or without contrast enhancement, in order to verify and quantify their presence and to correlate their number, morphology and location with the degree of disability, the clinical course, the evolution of the disease and the laboratory data, evaluating in each case the extent of demyelination and remyelination process and the degree of activation of innate immunity. The data obtained will be processed and evaluated to identify MRI and PET differences in the various disease courses and to obtain information on the different desease development paths in patients.

Study design Enrolled patients will undergo a brain MRI, a brain PET scan with amyloid tracer and functional assessment scales at the time of recruitment.

All patients will undergo clinical evaluation and various tests:

* EDSS and MS Functional Composite Scale
* Mini-BESTest
* TUG test, MSWS-12, Berg Balance Scale (BBS)
* The nine hole peg test (9-HPT) for right and left upper limb.
* Cognitive functions assessed by Brief International Cognitive Assessment for MS (BICAMS) and MMSE

Laboratory analysis of serum markers will be performed. Specifically, neuronal and glial cytoskeletal proteins (e.g. Nf-L, pN-FH, GFAP) as brain damage indices (axonal and cellular damage), will be considered and quantified.

The levels of specific neurotrophic factors (e.g. BDNF, GDNF) and cytokines (e.g. TNFα, IL-6, IL-1β, interferon) will be determined; there is evidence of their involvement in synaptic plasticity, cognitive and motor functions, and in the neuroinflammatory processes typical of MS.

MRI protocol Examinations will be performed on a 3T MRI scanner using a 32-channel head coil with sequences optimised and harmonised by the IRCCS Neuroscience Network.

The sequences that will be acquired will be:

1. T1-weighted sagittal volumetric image (MP-RAGE, 1 mm resolution) to study the morphology and encephalon volumetry
2. T2-FLAIR weighted sagittal volumetric image (1 mm resolution) for lesion localisation and contouring
3. a sequence of diffusion-weighted images (EPI, 2.5 mm resolution, b=1000 and 2000 s/mm2, 30 directions per shell) for the study of tissue microstructure and for the identification of pathology-relevant white matter bundles by tractography
4. a 3D multi-echo gradient echo sequence for quantitative susceptibility mapping (1 mm resolution, 8 echoes) for the study of local susceptibility
5. an fMRI resting-state sequence (EPI, 3 mm resolution, 200 volumes with a temporal resolution of 2.4 s) for the study of functional resting state networks.

PET protocol

The PET/CT study will be performed using a dual time acquisition protocol:

- Early acquisition Early acquisition starts with the patient already positioned on the PET/CT bed and venous access available.

A low-dose CT scan is performed for attenuation correction, the PET acquisition is started in list mode and a couple of seconds after the start, 300 MBq of 18F-Florbetaben is administered followed by washing with 10 ml of saline.

Early acquisition will last 30 minutes.

- Late acquisition A low-dose CT scan is performed to correct for attenuation and anatomical localisation, followed by a 20-minute list mode PET acquisition so that images are acquired after 90 minutes (tolerance: +10 minutes) of radiopharmaceutical uptake.

All PET reconstructions will have the following characteristics:

* 256 x 256 matrix, FOV 30 cm
* 3D-OSEM reconstruction algorithm with TOF and PSF and with standard corrections for decay, attenuation, scatter, dead time
* 8 iterations, 32 subsets, Gaussian filter with FWHM of 5 mm. Raw data will be available for possible different iterations, decided a posteriori, to improve image quality.

Patients do not need to be fasting or suspending current therapies.

MRI and PET evaluations MRI

1. Automated encephalic morpho-volumetric study (Freesurfer), by acquisition of conventional sequences (T2w, FLAIR 3D, T1w-3D), harmonised according to RIN protocol:

   1. cortical thickness;
   2. global brain atrophy;
   3. lesions burden;
   4. Normal-Appearing White Matter (NAWM).
2. Detection and study of chronic "smoldering" lesions using the QSM technique, which allows both qualitative and quantitative assessments of the extent of intralesional iron accumulation:

   1. Qualitative assessment:

      * Identification of Rim+ lesions, defined as "non-enhancing lesions with hyperintense perilesional rim", with iso-ipointense core;
      * Calculation of the global volume of Rim+ lesions (in mm3), with subsequent separate measurement of core and Rim.
   2. Quantitative assessment

      * calculation of the global susceptibility of the Rim+ lesions (expressed in ppb: parts per billion), compared to the CSF reference value;
      * calculation of susceptibility of Rim and core, separately.
3. Active lesions evaluation by assessing:

   1. Number of lesions showing contrastographic enhancement (qualitative assessment);
   2. Type of enhancement (nodular or shell-enhancement). The various parameters will be evaluated by three operators (radiologists with expertise in neuroradiology), with consensus agreement and a double check at 4 months after the first evaluation.

PET A slightly abbreviated protocol will be used with a 30-minute dynamic acquisition immediately after the injection of 18F-Florbetaben followed by a 20-minute delayed acquisition (this performed between 90 and 110 minutes after injection). The tracer binds to NAWM and in minor extent to the actively demyelinating plaques, which will be quantified. In addition, a semi-quantitative objective methodology will be used to obtain data on the degree of demyelination of the different cases examined by comparison of the data of the region of interest under investigation with NAWM uptake and a reference area uptake.

In particular, the semi-quantification foreseen is a SUVr where the uptake ROIs are the lesions pre-segmented by the neuroradiologist on MRI (FLAIR and T1 sequences), while for the reference ROIs several possibilities will be evaluated: the contralateral uptake ROIs (i.e. in the white matter if apparently normal on MRI), the white matter hot-spots in the late acquisition, the white matter average with the exclusion of the uptake ROIs. The dynamic uptake profile from the early acquisition will also be assessed, using different temporal reconstructions.

This semi-quantitative evaluation will be carried out in collaboration with colleagues from Nuclear Medicine and the National Institute of Nuclear Physics in Genoa, who have extensive experience in the field and have recently published semi-quantitative methods for the evaluation of PET investigation in Alzheimer's disease.

Sample size

This is an exploratory study of correlation between clinical, laboratory, MRI and PET findings. Considerations on sample size are omitted in the current study and may be included and perfectionated in future confirmatory studies.

Expected results The main objective of the study will be to verify the presence of correlations between PET and MRI images indicative of chronic inflammatory activity (smoldering plaques), of apparent absence of inflammatory activity (silent plaques without microglial Rim) or indicative of more recent inflammatory activity, in contrast-enhancing areas or in T2/Flair positive areas of not distant onset.

PET data will be correlated with conventional MRI parameters, and with clinical and laboratory data. The finding of significant correlations would support the role of PET as a useful tool for evaluating demyelination and remyelination activity, which may be characteristic of a certain disease phase or even possibly of specific types of individual patients.

Particular attention will be paid to study chronic lesions considering the promising results reported in recent studies showing the possibility to distinguish silent lesions from active chronic lesions (termed "smoldering") characterised by a core of complete demyelination and a periphery with activated microglial/macrophage elements.

The presence of this 'peripheral rim' can be quantitatively assessed in vivo by QSM (Quantitative Susceptibility Mapping) magnetic resonance sequences with 3T magnetic field study with good reliability compared to the histological correlate.

The association and fusion of structural MRI imaging data (related to both areas of demyelination and iron deposits) with PET data (related to amyloid deposits) may better allow to identify, within a cohort of patients with chronic demyelinating lesions, smoldering type lesions where demyelination process is still in progress and which therefore, in addition to indicating a predictive factor for the failure of the remyelination process, correlate with a longer duration of the disease and a more progressive course.

Dosimetry PET/CT examination with 18F-Florbetaben is justified in view of the risk/benefit ratio for the patient. Following administration of the radiopharmaceutical, the patient will inevitably receive a certain dose of radiation. The activity to be administered was set at 300 MBq, which is below the upper limit of 360 MBq, in order to obtain a PET examination of good diagnostic accuracy with a reasonable radiation dose.

ELIGIBILITY:
Inclusion Criteria:

* progressive stage of multiple sclerosis (both secondary and primary, SMP)
* patients in relapsing-remitting multiple sclerosis (RRMS)

Exclusion Criteria:

* a disability greater than 7
* patients with a cognitive impairment interfering with full study participation (Minimental score less than 24)
* patients with internal medical problems that in the opinion of the investigator may interfere with full participation and collaboration
* inability to undergo MRI or PET examinations
* ongoing pregnancy and lactation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
PET outcome | this evaluation is performed at the time of recruitment
  The main endpoint is to differentiate PET outcome in progressive forms compared to relapsing-remitting forms. It is expected that in RRMS forms, the degree of demyelination and of remyelination is lower and higher, respectively, than in progressive forms.

SECONDARY OUTCOMES:
correlation between PET data and MRI images and degree of disability | this evaluation is performed at the time of recruitment
  * Correlations between "smoldering plaques" identified on MRI and their degree of demyelination and remyelination detected on amyloid PET (Relationship between global susceptibility of Rim+ lesions and semi-quantitative data of tracer uptake in the region of interest)
  * Correlations between T2/Flair positive plaques and degrees of demyelination and remyelination
  * Relationship between number and extent of smoldering plaques and degree of disability
  * Relationship between extent of demyelination detected by amyloid PET and disability
  * Relationship between extent of remyelination detected by PET and disability
  * Relation between axonal damage found by laboratory tests (neurofilaments) and the presence of pro-inflammatory cytokines and MRI evidence of axonal impairment (atrophy); activation of innate immunity (microglial rem); presence of demyelination and remyelination at PET

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Trifirò, MD, Principal Investigator — ICS Maugeri Spa SB IRCCS
Locations (1):
- ICS Maugeri SpA SB IRCCS, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Absinta M, Sati P, Masuzzo F, Nair G, Sethi V, Kolb H, Ohayon J, Wu T, Cortese ICM, Reich DS. Association of Chronic Active Multiple Sclerosis Lesions With Disability In Vivo. JAMA Neurol. 2019 Dec 1;76(12):1474-1483. doi: 10.1001/jamaneurol.2019.2399. PMID 31403674
- [Background] Maggi P, Sati P, Nair G, Cortese ICM, Jacobson S, Smith BR, Nath A, Ohayon J, van Pesch V, Perrotta G, Pot C, Theaudin M, Martinelli V, Scotti R, Wu T, Du Pasquier R, Calabresi PA, Filippi M, Reich DS, Absinta M. Paramagnetic Rim Lesions are Specific to Multiple Sclerosis: An International Multicenter 3T MRI Study. Ann Neurol. 2020 Nov;88(5):1034-1042. doi: 10.1002/ana.25877. Epub 2020 Sep 9. PMID 32799417
- [Background] Absinta M, Lassmann H, Trapp BD. Mechanisms underlying progression in multiple sclerosis. Curr Opin Neurol. 2020 Jun;33(3):277-285. doi: 10.1097/WCO.0000000000000818. PMID 32324705
- [Background] Bagnato F, Gauthier SA, Laule C, Moore GRW, Bove R, Cai Z, Cohen-Adad J, Harrison DM, Klawiter EC, Morrow SA, Oz G, Rooney WD, Smith SA, Calabresi PA, Henry RG, Oh J, Ontaneda D, Pelletier D, Reich DS, Shinohara RT, Sicotte NL; NAIMS Cooperative. Imaging Mechanisms of Disease Progression in Multiple Sclerosis: Beyond Brain Atrophy. J Neuroimaging. 2020 May;30(3):251-266. doi: 10.1111/jon.12700. PMID 32418324
- [Background] Stankoff B, Poirion E, Tonietto M, Bodini B. Exploring the heterogeneity of MS lesions using positron emission tomography: a reappraisal of their contribution to disability. Brain Pathol. 2018 Sep;28(5):723-734. doi: 10.1111/bpa.12641. PMID 30020560
- [Background] Bodini B, Stankoff B. PET is necessary to make the next step forward in understanding MS pathophysiology - Yes. Mult Scler. 2019 Jul;25(8):1086-1087. doi: 10.1177/1352458519828298. Epub 2019 Feb 27. No abstract available. PMID 30810071
- [Background] Hogel H, Rissanen E, Vuorimaa A, Airas L. Positron emission tomography imaging in evaluation of MS pathology in vivo. Mult Scler. 2018 Oct;24(11):1399-1412. doi: 10.1177/1352458518791680. Epub 2018 Aug 9. PMID 30091657
- [Background] Calvi A, Haider L, Prados F, Tur C, Chard D, Barkhof F. In vivo imaging of chronic active lesions in multiple sclerosis. Mult Scler. 2022 Apr;28(5):683-690. doi: 10.1177/1352458520958589. Epub 2020 Sep 23. PMID 32965168
- [Background] Chen MK, Mecca AP, Naganawa M, Finnema SJ, Toyonaga T, Lin SF, Najafzadeh S, Ropchan J, Lu Y, McDonald JW, Michalak HR, Nabulsi NB, Arnsten AFT, Huang Y, Carson RE, van Dyck CH. Assessing Synaptic Density in Alzheimer Disease With Synaptic Vesicle Glycoprotein 2A Positron Emission Tomographic Imaging. JAMA Neurol. 2018 Oct 1;75(10):1215-1224. doi: 10.1001/jamaneurol.2018.1836. PMID 30014145
- [Background] Chincarini A, Peira E, Morbelli S, Pardini M, Bauckneht M, Arbizu J, Castelo-Branco M, Busing KA, de Mendonca A, Didic M, Dottorini M, Engelborghs S, Ferrarese C, Frisoni GB, Garibotto V, Guedj E, Hausner L, Hugon J, Verhaeghe J, Mecocci P, Musarra M, Queneau M, Riverol M, Santana I, Guerra UP, Nobili F. Semi-quantification and grading of amyloid PET: A project of the European Alzheimer's Disease Consortium (EADC). Neuroimage Clin. 2019;23:101846. doi: 10.1016/j.nicl.2019.101846. Epub 2019 May 4. PMID 31077984
- [Background] Bodini B, Veronese M, Garcia-Lorenzo D, Battaglini M, Poirion E, Chardain A, Freeman L, Louapre C, Tchikviladze M, Papeix C, Dolle F, Zalc B, Lubetzki C, Bottlaender M, Turkheimer F, Stankoff B. Dynamic Imaging of Individual Remyelination Profiles in Multiple Sclerosis. Ann Neurol. 2016 May;79(5):726-738. doi: 10.1002/ana.24620. PMID 26891452
- [Background] Kaunzner UW, Kang Y, Zhang S, Morris E, Yao Y, Pandya S, Hurtado Rua SM, Park C, Gillen KM, Nguyen TD, Wang Y, Pitt D, Gauthier SA. Quantitative susceptibility mapping identifies inflammation in a subset of chronic multiple sclerosis lesions. Brain. 2019 Jan 1;142(1):133-145. doi: 10.1093/brain/awy296. PMID 30561514
- [Background] Mehta V, Pei W, Yang G, Li S, Swamy E, Boster A, Schmalbrock P, Pitt D. Iron is a sensitive biomarker for inflammation in multiple sclerosis lesions. PLoS One. 2013;8(3):e57573. doi: 10.1371/journal.pone.0057573. Epub 2013 Mar 14. PMID 23516409
- [Background] Absinta M, Sati P, Fechner A, Schindler MK, Nair G, Reich DS. Identification of Chronic Active Multiple Sclerosis Lesions on 3T MRI. AJNR Am J Neuroradiol. 2018 Jul;39(7):1233-1238. doi: 10.3174/ajnr.A5660. Epub 2018 May 3. PMID 29724768
- See also: Radiation exposure by [F18]Florbetaben, a new PET tracer for detection of cerebral β-amyloid in Caucasian and Asian healthy volunteers — https://jnm.snmjournals.org/content/51/supplement_2/1448